CLINICAL TRIAL: NCT00487825
Title: A 26-week, Phase II, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Assess the Response to Treatment (ACR50) and to Determine a Biomarker Profile in Responders to ACZ885 (Anti-interleukin-1beta Monoclonal Antibody) Plus MTX as Compared to MTX Alone in Early Rheumatoid Arthritis Patients
Brief Title: Safety and Efficacy of Intravenous ACZ885 and Oral Methotrexate Therapy in Patients With Early Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885A2204
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Rheumatoid Arthritis
Keywords: ACR20, ACR50, ACZ885 (anti-interleukin-1beta monoclonal antibody), rheumatoid arthritis, methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — canakinumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canakinumab + Methotrexate (Experimental): Canakinumab, human anti-interleukin-1beta monoclonal antibody plus Methotrexate (MTX). Intravenous (IV) Infusion of 600mg canakinumab on Day 1, 15 continuing every 4 weeks up to week 26. MTX was given as variable dosing regimen of 7.5 mg-15 mg weekly.
  Interventions: Drug: Canakinumab (investigational); Drug: Methotrexate (MTX)
- Methotrexate + placebo (Active Comparator): Methotrexate (MTX) was given as variable dosing regimen of 7.5 mg-15 mg weekly. Intravenous (IV) Placebo Solution, given in the same mode of administration as the canakinumab solution.
  Interventions: Drug: Placebo; Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Canakinumab (investigational) — Canakinumab was supplied in 6 mL colorless glass vials each containing nominally 150 mg canakinumab (with 20% overfill). The vials were kept at 2-8°C. At the investigator's site, solutions for infusion were prepared depending on the volume and dose administered.
  Other Names: ACZ885
  Arms: Canakinumab + Methotrexate
Drug: Placebo — Matching placebo was supplied in form of a lyophilized cake (Powder for Solution for Infusion). At the investigator's site, solutions for infusion were prepared depending on the volume and dose administered.
  Arms: Methotrexate + placebo
Drug: Methotrexate (MTX) — Methotrexate (MTX) was supplied in tablet form, each of 2.5 mg strength.

SUMMARY:
This study was intended to evaluate the safety and efficacy of intravenous (IV) ACZ885 and oral methotrexate (MTX) therapy in patients with early rheumatoid arthritis (RA)

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of 18 to 75 years of age (inclusive)
* Recent definite diagnosis of rheumatoid arthritis (RA) (<3 years since diagnosis), classified by American Rheumatism Association 1987 revised criteria.
* Candidate for methotrexate (MTX) or biologic due to erosive arthritis, with no contraindications to such therapy, including:
* Negative tuberculin skin test reaction
* Normal chest X-ray (within the last year) prior to possibility of receiving MTX (r/o lung fibrosis).
* Active disease: at least 6 swollen and 6 painful tender joints of 28 joint count,
* Vital signs should be within the following ranges:
* 18-59 years of age: oral temperature between 35.0-37.5 °C systolic blood pressure, 90-140 mm Hg diastolic blood pressure, 50-90 mm Hg pulse rate, 40 - 90 beats per minute
* 60-75 years of age: oral temperature between 35.0-37.5 °C systolic blood pressure, 100-160 mm Hg diastolic blood pressure, 50-100 mm Hg pulse rate, 50 - 100 beats per minute
* Women of child-bearing potential willing to practice double-barrier contraception during the study for at least 3 months following last study drug administration. Postmenopausal women must have no regular menstrual bleeding for at least 1 year prior to inclusion. Surgically sterilized women at least 6 months prior to screening.

Male patients must be using a double-barrier local contraception and refrain from fathering a child in the 3 months following last study drug administration.

* Weight: at least 45 kg; body mass index (BMI) within the range of 18 to 34.
* Oral corticosteroids are permitted as long as patients are on a stable dose (up to 10 mg) for at least 4 weeks before study start.

Exclusion Criteria:

* Unable to have Magnetic Resonance Imaging (MRI) of wrist.
* Patients with magnetizable metal parts/devices on and in the body that could interfere with the MRI
* Patients with an unstable active medical condition that could impair evaluation of study results.
* Previous treatment with biological therapy or MTX.
* Limited kidney function (creatinine clearance under 60 ml/min)
* Previous treatment with other disease-modifying anti-rheumatic drugs such as sulfasalazine, hydroxychloroquine within 4 weeks of screening.
* Corticosteroids injections into joints within 4 weeks prior to screening.
* Participation in any clinical investigation within 4 weeks prior to study start or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Blood donation or loss of > 400 mL within 8 weeks before study start, or longer if required by local regulation.
* Significant illness within 2 weeks of study start.
* Past personal or family medical history of clinically significant ECG abnormalities or cardiac issues.
* History of:

  * fainting, orthostatic hypotension, sinus arrhythmia asthma and chronic obstructive pulmonary disease, clinically significant drug allergy or urticaria, eczematous dermatitis, and/or known hypersensitivity to the study drug or drugs similar to the study drug.
  * disease of the blood building system, serious or active infections, gastric ulcers.
  * surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the patient in case of participation in the study.
  * immunodeficiency diseases, including a positive Human Immunodeficiency Virus (HIV) (ELISA and Western blot) test result.
  * positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
  * drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (22):
- United States (17):
  - Rheumatology Associates of Northern Alabama (Dr. William Shergy), Huntsville, Alabama
  - Clinic for Rheumatic Diseases (Dr. Richard Jones, III), Tuscaloosa, Alabama
  - Arizona Arthritis and Rheumatology Research (Dr. Paul Caldron), Paradise Valley, Arizona
  - Jacksonville Center for Clinical Research (Dr. Steven Mathews), Jacksonville, Florida
  - Center for Arthritis and Rheumatic Diseases (Dr. Michael Weitz), South Miami, Florida
  - West Broward Rheumatology Associates, Incorporated (Dr. Elias Halpert), Tamarac, Florida
  - Rockford Orthopedic Associates (Dr. Richard Olson), Rockford, Illinois
  - Mercy Arthritis and Osteoporosis Center (Dr. Alan Braun), Urbandale, Iowa
  - Clayton Medical Research (Dr. Iri Don), Richmond Heights, Missouri
  - Westroads Medical Group (Dr. William Palmer), Omaha, Nebraska
  - Arthritis Center of Reno (Dr. Malin Prupas), Reno, Nevada
  - Oklahoma Center for Arthritis therapy and Research (Dr. James McKay), Tulsa, Oklahoma
  - MetaClin Research, Incorporated (Dr. Paul Pickrell), Austin, Texas
  - John M. Joseph, MD (Dr. John Joseph), Carlton, Texas
  - Southwest Rheumatology, P.A. (Dr. Atul Singhal), Mesquite, Texas
  - Arthritis Clinic of Northern Virginia (Dr. Philip Kempf), Arlington, Virginia
  - Arthritis Northwest Rheumatology, PLLC (Dr. Jeffrey Butler), Spokane, Washington
- Novartis Investigative site, Brussels, Belgium
- Novartis investigative site, Nuremberg, Germany
- Novartis investigative site, Milan, Italy
- Novartis Investigative site, Arnhem, Netherlands
- Novartis investigative site, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A 26-week, phase II, multi-center, randomized, double-blind, placebo-controlled study to assess the response to treatment and to determine a biomarker profile in responders to Canakinumab plus MTX as com-pared to MTX alone in early rheumatoid arthritis patients. Study starting 16-Mar 2007 and ending 19 Dec 2008.
Groups:
- Canakinumab + Methotrexate: Canakinumab, human anti-interleukin-1beta monoclonal antibody plus Methotrexate (MTX). Intravenous (IV) Infusion of 600mg canakinumab on Day 1, 15 continuing every 4 weeks up to week 26. Methotrexate is given as variable dosing regimen of 7.5 mg-15 mg weekly.
- Methotrexate: Methotrexate is given as variable dosing regimen of 7.5 mg-15 mg weekly. Intravenous (IV) Placebo Solution, given in the same mode of administration as the canakinumab solution.
Period: Overall Study
Arm/Group | Canakinumab + Methotrexate | Methotrexate
Started | 52 ("Started" indicates Intent-to-treat population (ITT)) | 26
Completed | 46 | 21
Not Completed | 6 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Other | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab + Methotrexate | Methotrexate | Total
Number analyzed (Participants) | 52 | 26 | 78
Age Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (12.78) | 49.7 (14.15) | 50.9 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 18 | 63
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Response to Intravenous Canakinumab and Oral Methotrexate (MTX) Compared to MTX Alone as Determined by 50% Improvement in Symptoms According to the American College of Rheumatology Criteria (ACR50)
Description: A patient was considered as improved according to the ACR50 criteria if she/he had at least a 50 % improvement in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures:
  * Patient's pain assessment (Visual Analogue Scale (VAS) 100 mm)
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score)
  * Acute phase reactant (high sensitivity C-reactive Protein (hsCRP))
Time Frame: 6, 14, and 26 weeks of treatment
Population: Intent-to-treat population (ITT)
Measure: Number; unit: Participants
Arm/Group | Canakinumab + Methotrexate | Methotrexate
Number analyzed (Participants) | 52 | 26
Participants
  ACR50 6 weeks after first dosing | 10 | 5
  ACR50 14 weeks after first dosing | 19 | 9
  ACR50 26 weeks after first dosing | 24 | 11

2. Secondary Outcome: Response to Intravenous (IV) Canakinumab and Oral Methotrexate (MTX) Therapy (ACR20, 70, 90) Compared to MTX Alone
Description: A patient was considered as improved according to the criteria of ACR 20 equaling at least 20%, ACR70 = 70%, and ACR90 = 90% improvement in the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures:
  * Patient's pain assessment (Visual Analogue Scale (VAS) 100 mm)
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score)
  * Acute phase reactant (high sensitivity C-reactive Protein (hsCRP))
Time Frame: At 6 weeks, 14 weeks, and 26 weeks
Population: Intent-to-treat population (ITT)
Measure: Number; unit: Participants
Arm/Group | Canakinumab + Methotrexate | Methotrexate
Number analyzed (Participants) | 52 | 26
Participants
  ACR20 6 weeks after first dosing | 32 | 13
  ACR20 14 weeks after first dosing | 38 | 16
  ACR20 26 weeks after first dosing | 39 | 20
  ACR70 6 weeks after first dosing | 1 | 3
  ACR70 14 weeks after first dosing | 6 | 3
  ACR70 26 weeks after first dosing | 17 | 9
  ACR90 6 weeks after first dosing | 0 | 0
  ACR90 14 weeks after first dosing | 1 | 0
  ACR90 26 weeks after first dosing | 4 | 2

3. Secondary Outcome: Percentage of Participants Achieving a Good European League Against Rheumatism (EULAR) Response (Based on the Disease Activity Score (DAS28)) at 26 Weeks
Description: At each visit (including baseline) the DAS28 is derived as: DAS28 = 0.56*√ (tender28) + 0.28 * √ (swollen28) + 0.36 * loge(CRP+1) + 0.014*PGDA+ 0.96; where tender28 is the tender 28-joint count, swollen28 is the swollen 28-joint count, PGDA is the patient's global assessment of disease activity. Patients can be scored on a range of 0 to 10. When current DAS < 3.2, good response is defined as >1.2 improvement in DAS from baseline and non-response is improvement of ≤0.6. When current DAS >5.1, non-response is improvement of >0.6 but ≤1.2 . All others are moderate responses.
Time Frame: At 26 weeks
Population: Intention to treat (ITT) population
Measure: Number; unit: Percentage of Participants
Arm/Group | Canakinumab + Methotrexate | Methotrexate
Number analyzed (Participants) | 52 | 26
Percentage of Participants
  Good responders | 46.2 | 30.8
  Mild responders | 28.8 | 42.3
  Non responders | 17.3 | 11.5

4. Secondary Outcome: The Number of Participants in Clinical Remission Based on Disease Activity Score (DAS)28 and Simplified Disease Activity Index (SDAI)
Description: At each visit (including baseline) the DAS28 and SDAI variables were derived using the following formulas:
  DAS28 = 0.56*√ (tender28) + 0.28 * √ (swollen28) + 0.36 * loge(CRP+1) + 0.014*PGDA+ 0.96; SDAI = tender28 + swollen28 + CRP + (PGDA / 10) + (EGDA / 10) where tender28 is the tender 28-joint count, swollen28 is the swollen 28-joint count, CRP is C-reactive protein, PGDA is the patient's global assessment of disease activity and EGDA is the physician's global assessment of disease activity.
  The Number of Participants in clinical remission is defined as the DAS28 ≤ 2.6 or SDAI ≤ 3.3.
Time Frame: At 6 weeks, 14 weeks and 24 weeks
Population: Intention to treat (ITT) population
Measure: Number; unit: Participants
Arm/Group | Canakinumab + Methotrexate | Methotrexate
Number analyzed (Participants) | 52 | 26
Participants
  After 6 weeks | 6 | 3
  After 14 weeks | 13 | 3
  After 26 weeks | 20 | 6

ADVERSE EVENTS:
Time Frame: 26 weeks plus a follow-up period of 3 months
Arm/Group | Canakinumab + Methotrexate | Methotrexate
Serious Adverse Events (participants affected / at risk) | 1/52 | 2/26
Other Adverse Events (participants affected / at risk) | 36/52 | 21/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab + Methotrexate (N=52) | Methotrexate (N=26)
Lip oedema (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab + Methotrexate (N=52) | Methotrexate (N=26)
Vertigo (Ear and labyrinth disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 8 | 9
Vomiting (Gastrointestinal disorders) | 4 | 3
Fatigue (General disorders) | 7 | 2
Nodule (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 4 | 2
Bronchitis (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 6 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Dizziness (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 7 | 2
Depression (Psychiatric disorders) | 3 | 2
Sleep disorder (Psychiatric disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Hypertension (Vascular disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.